CLINICAL TRIAL: NCT00715819
Title: Use of Otoscope as a Non-invasive Tool for Diagnosis of Pilomatricoma
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: SU-07092008-1245; eProtocol #:13219
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pilomatrixoma
MeSH Terms: conditions — Pilomatrixoma

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Stanford University Dermatology Clinics and Lucile Packard Children's Hospital are evaluating the use of the otoscope for the diagnosis of skin lesions. We are particularly looking for children and/or adults with nodules, cysts, tumors, or pilomatricomas. The study will take 15-30 minutes and we will use light to examine and take a picture of your skin lesion. There is no monetary compensation for participating in the study.

DETAILED DESCRIPTION:
Pilomatricoma is a benign tumor that presents as a 3-30mm firm, solitary, deep dermal or subcutaneous tumor on the head, neck, or upper extremities. The clinical diagnosis is often made by the firm, sometimes rock hard texture of the skin. The diagnosis can be confirmed by a skin biopsy and/or excision of the lesion. We have recently noted that pilomatricomas appear as a black mass in the skin when the lesion is transilluminated by placing the light of a fiberoptic otoscope adjacent to the skin lesion. We would like to confirm our impression by a prospective study using transillumination to examine subcutaneous tumors in the skin. Pilomatricoma is also known as a benign calcifying or calcified epithelioma, pilomatrixoma, or a calcifying epithelioma of Malherbe.

ELIGIBILITY:
Inclusion Criteria:- Potential participants will be any patient that is seen at Stanford Dermatology or LPCH that has a cyst, nodule, vesicle, tumor, or possible pilomatricoma Exclusion Criteria:- Inability of subject or subject's guardian to understand informed consent form.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Odmara Liz Barreto-Chang, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States